CLINICAL TRIAL: NCT00786773
Title: Epidemiological Survey to Describe Impact of Reflux Disease on Everyday Life in GERD Patients Before and After 4 Weeks Treatment
Brief Title: Survey to Describe Impact of Reflux Disease on Everyday Life in GERD Patients Before and After 4 Weeks Treatment.
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Le Van Phuc, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-GVN-DUM-2008/1
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; reflux symptom; heartburn; acid regurgitation; PPI; H2RA; antacid
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: GERD patients who will be treated for GERD with PPI, H2RA, antacid, prokinetics, combination therapy

SUMMARY:
To describe the change of impact of reflux symptoms on the everyday life perceived by patients before and after 4 weeks treatment by using GERD Impact Scale questionnaire (GIS) by total GERD patient population and by treatment group; and to describe the concordance between patient-reported and physician-reported symptom load.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GERD diagnosed clinically or by endoscopy and prescribed with medical treatments
* Provision of written informed consent

Exclusion Criteria:

* Patients cannot read and/or understand GIS
* Patients with the history or symptoms of peptic ulcer, gastrointestinal cancer, serious or malignant diseases (anorexia, weight loss, anemia, fever …)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target survey population is existing GERD patients or newly diagnosed GERD patients, who will be treated for GERD with PPI, H2RA, antacid, prokinetics, combination therapy ... at Visit 1 and will come back after 4 weeks for clinical re-assessment (Visit 2)
Sampling Method: Probability Sample
Enrollment: 2091 (Actual)
Dates: Start 2008-10; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Type, frequency and severity of the GERD symptoms | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ta Long, Principal Investigator — Vietnam Association of Gastroenterology; Dao Van Long, Principal Investigator — Medical University of Hanoi; Tran Kieu Mien, Principal Investigator — HCMC Association of Gastroenterology; Le Thanh Ly, Principal Investigator — Cho Ray Hospital
Locations (18):
- Vietnam (18):
  - Research Site, Long Xuyen, An Giang
  - Research Site, Qui Nhon, Binh Dinh
  - Research Site, Buon Ma Thuot, Dac Lac
  - Research Site, Biên Hòa, Dong Nai
  - Research Site, Thống Nhất, Dong Nai
  - Research Site, Cao Lanh, Dong Thap
  - Research Site, Sa Dec, Dong Thap
  - Research Site, Nha Trang, Khanh Hoa
  - Research Site, Huế, Thừa Thiên Huế Province
  - Research Site, Can Tho
  - Research Site, Cà Mau
  - Research Site, Da Nang
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Mỹ Tho
  - Research Site, Nam Định
  - Research Site, Thái Bình